CLINICAL TRIAL: NCT01976013
Title: Prediction of Major Bleeding in Extremely Low Birth Weight Infants (<1000g) by Sequential Coagulation Monitoring
Brief Title: Prediction of Major Bleeding in ELBW-infants (<1000g) by Sequential Coagulation Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoc.Prof.MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUV-Coagu
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Intraventricular Haemorrhage; Pulmonary Haemorrhage
Keywords: PT; INR; intraventricular haemorrhage; pulmonary haemorrhage; ELBW infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coaguchek (Other): infants will receive sequential coagulation checks
  Interventions: Device: Coaguchek

INTERVENTIONS:
Device: Coaguchek — The investigators plan to draw 10μL blood (i.e. approximately 1/5000 of the blood volume of an ELBW infant) within the scope of routine blood sampling. Thus, the number of blood samples will be variable. A cumulative sample volume for the whole study period will not exceed 300μL.

SUMMARY:
Up to now, only data about early and single coagulation screening exist in extreme low birth weight infants (ELBW) infants. In neonatal practice, coagulation abnormality in preterm babies is primarily investigated by measuring prothrombin time (PT). In fact, FVII activity, which is an important determinant of PT, is strongly associated with bleeding risk. Thus, a method to measure PT with small volume samples (10μL) provides the possibility for serial monitoring even in ELBW infants (CoaguChek®XS, Roche Diagnostics, Vienna, Austria)). Substitution of fesh frozen plasma seemed beneficial in ELBW infants and first trials with rFVII revealed promising results in this patient population. Thus, coagulation monitoring might lead to early and adequate therapy and therefore to a better outcome. The investigators hypothesize that ELBW infants (<1000g birth weight) with primary severe prolongation of prothrombin time or development of severe prothrombin prolongation during sequential monitoring may have more frequent and more severe bleeding incidents (Intraventricular haemorrhage and pulmonary haemorrhage). The investigators aim to explore whether monitoring of PT can predict bleeding events in ELBW children.

DETAILED DESCRIPTION:
It was recently reported that "early", i.e. in the first 48h of life, coagulation screening may identify infants at risk of severe IVH. Unfortunately, in the past screening for coagulation abnormalities and correction of haemostatic defects by prothrombin complex concentrate, cryoprecipitate or platelet concentrates) and fresh frozen plasma (FFP) had limited effects in preterm infants. This could have been due to the short duration of action, incomplete restoration of coagulation or the water and osmotic load associated with FFP administration. However recently, using a coagulopathy screening strategy (one blood sample within the first 2h after birth) and substitution with FFP decreased the risk of developing IVH in infants born at 23 to 26 weeks of gestation. Recombinant Factor VII (rFVII) provides a new therapeutic option to overcome FFP associated side effects. Small trials, including infants with pulmonary hemorrhage, showed the safety and effectiveness of rFVII in VLBW infants; however no randomised controlled trials have been published so far. As outlined above, bleeding complications are still a major problem in extremely low birth weight (ELBW) infants and coagulation abnormalities are associated with bleeding. Up to now, only data about early and single screening exist and coagulation monitoring with multiple blood sampling was not applied.

In neonatal practice, coagulation abnormality in preterm babies is primarily investigated by measuring prothrombin time (PT). In fact, FVII activity, which is an important determinant of PT, is strongly associated with bleeding risk. Thus, a method to measure PT with small volume samples (10μL) provides the possibility for serial monitoring even in ELBW infants.

Substitution of FFP seemed beneficial in ELBW infants and first trials with rFVII revealed promising results in this patient population. Thus, coagulation monitoring might lead to early and adequate therapy and therefore to better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a birth weight <1000g
* signed informed consent

Exclusion Criteria:

* Congenital heart disease
* major congenital birth defects

Ages: 2 Minutes to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
major bleeding | 30 days
  pulmonary bleeding, intraventricular hemorrhage

SECONDARY OUTCOMES:
mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria